CLINICAL TRIAL: NCT07260799
Title: Clinical Performance of Capillary Blood Samples Collected Using the Tasso+ Serum Gel Capillary Blood Collection System for Clinical Chemistry Testing of 14 Analytes on an Abbott Alinity Analyzer
Status: Recruiting | Type: Observational
Sponsor: Tasso Inc. (Industry)
Collaborators: American Research Labs (Industry)
Responsible Party: Sponsor
Other Study IDs: T23-03
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Serum Analytes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Tasso+ Serum Gel Capillary Blood Collection System: Comparison of serum analyte results from capillary blood collected using the Tasso+ Serum Gel Capillary Blood Collection System vs. venous blood obtained via traditional venipuncture.
  Interventions: Diagnostic Test: Tasso+ Serum Gel Capillary Blood Collection System

INTERVENTIONS:
Diagnostic Test: Tasso+ Serum Gel Capillary Blood Collection System — Clinical evaluation of capillary blood samples collected using the Tasso+ Serum Gel Capillary Blood Collection System for downstream analyte testing.

SUMMARY:
The purpose of this single-visit study is to demonstrate the performance of capillary blood samples collected with the Tasso+ Serum Gel Capillary Blood Collection System compared to venous reference samples for downstream analyte testing at a clinical laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18-85 years with no previous experience with the Tasso+ lancet
2. Willing and able to provide written informed consent prior to study entry
3. Willing and able to adhere to study assessments, schedule, prohibitions and restrictions as described in the protocol
4. Healthy individuals or patients with abnormal analyte values (verified or likely to be) within intended clinical reference ranges as indicated by standard of care testing and/or past medical history, in the judgement of the investigator

Exclusion Criteria:

1. Present with abnormal skin integrity or atypical skin health near/on arm collection sites
2. Mental or physical impairment which would preclude participation in the judgement of the investigator or qualified designee
3. Trained clinical laboratory and healthcare personnel who have worked in the field in the previous 5 years
4. Any condition which, in the opinion of the investigator or delegate, makes the participant unsuitable for this study (including, but not limited to, any mental or physical impairment which would preclude provision of adequate and knowledgeable consent)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals or patients with abnormal analyte values (verified or likely to be) within intended clinical reference ranges as indicated by standard of care testing and/or past medical history.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Number participants for which there is statistical equivalence between serum biomarker results obtained from capillary blood vs. venous blood | 48 Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Celesta / American Research Labs, Atlantis, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Research results are proprietary; no sharing with other researchers is anticipated.